CLINICAL TRIAL: NCT03527784
Title: PRESTOMA- A Prospective Randomized Controlled Multicenter Trial Comparing Three Meshes for Prevention of Parastomal Hernia After Abdominoperineal Resection for Rectal Adenocarcinoma
Brief Title: Prestoma-Trial for Parastomal Hernia Prevention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Parastomal Parietex withdrawn from market by the manufacturer.
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Elisa Makarainen-Uhlback, M.D., University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 85/2018
Record Dates: First submitted 2018-05-02; First posted 2018-05-17 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Rectal Adenocarcinoma
Keywords: rectal adenocarcinoma; abdominoperineal resection; hernia prophylaxis
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Prestoma is a prospective randomized controlled multicenter trial.
Who Masked: Participant
Masking Description: Subject is blinded of the mesh used. Outcome at 12 month follow-up is assessed by surgeon who was not involved in the operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parietene Macro (Active Comparator): Parietene Macro is a macroporous synthetic mesh.
  Interventions: Device: Parietene Macro
- Parietex Parastomal (Active Comparator): Parietex Parastomal is a synthetic mesh with resorbable collagen lining to prevent attachments.
  Interventions: Device: Parietex Parastomal
- Dynamesh IPST (Active Comparator): Dynamesh IPST is synthetic mesh with central tube to accommodate bowel tightly designed to prevent and treat parastomal hernia.
  Interventions: Device: Dynamesh IPST

INTERVENTIONS:
Device: Parietene Macro — Parietene Macro is used on retromuscular sublay position. The bowel is brought through opening in the middle of the mesh.
  Arms: Parietene Macro
Device: Parietex Parastomal — Parietex Parastomal is used on intraperitoneal onlay position by modified Sugarbaker technique to prevent parastomal hernia.
  Arms: Parietex Parastomal
Device: Dynamesh IPST — Dynamesh IPST is used on intraperitoneal onlay position to prevent parastomal hernia
  Arms: Dynamesh IPST

SUMMARY:
Prestoma Trial is designed to compare the safety and efficiency of three different meshes and techniques to prevent parastomal hernia after laparoscopic or robotic-assisted abdominoperineal resection for rectal adenocarcinoma.

DETAILED DESCRIPTION:
Parastomal hernia after permanent colostomy formation is a common problem. The European Hernia Society recommends the use of prophylactic mesh when the stoma is constructed. So far, there're no trials comparing the methods to prevent the parastomal hernia.

Prestoma Trial is designed to compare the most researched retromuscular mesh (Parietene Macro by Medtronic) with two different types of intraperitoneal meshes (Parietex Parastomal by Medtronic and Dynamesh IPST) in parastomal hernia prevention after laparoscopic or robotic-assisted abdominoperineal resection for rectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Abdominoperineal resection for rectal cancer with permanent end colostomy, either by laparoscopic technique or robotic assistance
* 18 years or older
* Patient has a life expectancy of at least 12 months.
* Patient signs the Informed consent and agrees to attend all study visits.

Exclusion Criteria:

* Abdominoperineal resection by laparotomy or conversion to laparotomy
* Patient with a comorbid illness or condition that would preclude the use of surgery (ASA 4-5).
* Patients with concurrent or previous malignant tumors within 5 years before study enrollment
* Patients with T4b tumors which impose a multi-organ resection
* Rectal malignancy other than adenocarcinoma
* Potentially curable resection not possible
* Patient undergoing emergency procedures
* Planned rectal surgery along with major concomitant procedures (e.g. hepatectomies, other intestinal resections).
* Metastatic disease with life expectancy of less than 1 year
* Pregnant or suspected pregnancy
* Patients living geographically distant and/or unwilling to return for follow-ups or comply with all study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Incidence of parastomal hernia | 1 year
  The primary outcome is incidence of parastomal hernia at 12 months follow up, detected clinically or on CT scan.

SECONDARY OUTCOMES:
Surgical infections | 30 days
  Surgical infections due to primary surgery, defined by CDC (Centers for Disease Control) definition for surgical site infection.
Complications | 30 days
  The incidence of complications defined by Clavien-Dindo Classification
Stoma related complications | 5 years
  Any complications related to stoma
Reoperation rate | 5 years
  Reoperation needed for any reason related to previous surgery
Operative time | 30 days
  Total time needed in operation theatre and time needed for mesh application
Length of stay | 30 days
  Length of stay at the hospital.
Quality of Life measured by RAND 36 | 5 years
  Quality of life measured by The RAND 36-Item Health Survey 1.0 which assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions with a scale 0-100, higher the score, better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Mäkäräinen-Uhlbäck, M.D., Principal Investigator — Oulu University Hospital
Locations (6):
- Finland (6):
  - Helsinki University Hospital, Helsinki
  - Jyväskylä Central Hospital, Jyväskylä
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No